CLINICAL TRIAL: NCT02402231
Title: Explorative Open Phase II-study, Food Allergy Suppression Therapy During Protection With Xolair
Brief Title: Treatment of Severe Peanut Allergy With Xolair (Omalizumab) and Oral Immunotherapy
Acronym: FASTX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Caroline Nilsson (Other)
Responsible Party: Sponsor-Investigator, Caroline Nilsson, MD, PhD, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FASTXP2013; 2012-005625-78 (EudraCT Number)
Record Dates: First submitted 2013-11-28; First posted 2015-03-30 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omalizumab (Experimental): Omalizumab is given to protect the study object from severe allergic reactions while they are going through oral immunotherapy with peanuts. There wïll be only one arm. The study objects are their own controls by also having allergy to airborne allergens. The dose is calculated by the study objects body mass and number of total IgE antibodies.
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — Omalizumab is the treatment during oral immunotherapy with peanuts as protection

SUMMARY:
Severe peanut allergy is different from other allergic reactions because it can lead to fatal reactions and is an invisible disability. There is no cure today. The purpose of this study is to treat children and adolescents with severe peanut allergy with oral immunotherapy with peanuts under the protection of anti-IgE (immunoglobulin E) antibodies (omalizumab), and thereby inducing tolerance to peanuts. The treatment will be monitored by basophil cell stimulation (CD-sens).

DETAILED DESCRIPTION:
Oral immunotherapy (OIT), where the food protein is consumed in increasing amounts, have been studied with good results, but allergic reactions has been a major problem. Anti-IgE antibodies (omalizumab) block allergy antibodies so that the allergic reaction is absent. A new test in which basophil cells stimulated with allergen in vitro, CD-sens, showing cell sensitivity, correlates well to peanut challenges.

Twenty children/adolescents, 12 to 22 years, with severe peanut allergy will be treated with omalizumab and the effect evaluated with CD-sens. If the CD-sens is negative a peanut challenge will be performed. If the challenge is negative the OIT will start: 1, 2, 4, 8 g peanuts/day in two-week intervals followed by a maintenance dose of 10 g peanuts/day while continuing treatment with omalizumab. If the CD-sens is still negative the withdrawal of omalizumab will start by halving the dose in several steps.

The study is independent of pharmaceutical companies. Omalizumab is dosed according to body mass and the amount of total IgE antibodies and therefore every individual has an individual study duration. In average the duration of the study is estimated to 52 weeks +/-40/20 weeks. Inclusion in the study is expected to last for the 2 coming years.

A treatment without serious side effects for those with severe food allergies would give a great benefit with reduced anxiety and fear, but also major health economic benefits in the form of fewer hospitalizations, sick leave, and to a greater extent completed school and education.

ELIGIBILITY:
Inclusion Criteria:

* IgE to peanut, Ara h 1, Ara h 2 and Ara h 3
* IgE to an airborne allergen i.e. cat, dog, horse, birch, grass etc.
* Clinical allergic reactions to peanut the last 5 years
* Positive conjunctival challenge to the selected airborne allergen
* Positive CD-sens to peanut and the selected airborne allergen
* IgE according to the recommendations of the manufacturer
* Written consent

Exclusion Criteria:

* No severe diseases like renal failure, hart disease, immunodeficiency, diabetes or other severe chronic diseases
* Pregnancy
* No previous hypersensitivity reactions to sucrose, histidine, polysorbat 20 or omalizumab

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2013-10; Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Peanut challenge. The peanut challenge can be positive i.e. the study object reacts to peanuts with allergic symptoms or negative i.e. no reaction in two hours after completed challenge. | The participants will be followed for the duration of Xolair treatment and oral immunotherapy, an expected average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Nilsson, MD, PhD, Principal Investigator — Dept of Clinical Science and Education, Karolinska Institutet
Locations (1):
- Sachs´ Children´s Hospital, Södersjukhuset, Stockholm, Sweden

REFERENCES:
- [Derived] Bjorkander S, Merid SK, Brodin D, Brandstrom J, Fagerstrom-Billai F, van der Heiden M, Konradsen JR, Kabesch M, van Drunen CM, Golebski K, Maitland-van der Zee AH, Potocnik U, Vijverberg SJH, Nopp A, Nilsson C, Melen E. Transcriptome changes during peanut oral immunotherapy and omalizumab treatment. Pediatr Allergy Immunol. 2022 Jan;33(1):e13682. doi: 10.1111/pai.13682. Epub 2021 Oct 31. No abstract available. PMID 34669990
- [Derived] Brandstrom J, Vetander M, Sundqvist AC, Lilja G, Johansson SGO, Melen E, Sverremark-Ekstrom E, Nopp A, Nilsson C. Individually dosed omalizumab facilitates peanut oral immunotherapy in peanut allergic adolescents. Clin Exp Allergy. 2019 Oct;49(10):1328-1341. doi: 10.1111/cea.13469. Epub 2019 Aug 15. PMID 31329313
- [Derived] Brandstrom J, Vetander M, Lilja G, Johansson SG, Sundqvist AC, Kalm F, Nilsson C, Nopp A. Individually dosed omalizumab: an effective treatment for severe peanut allergy. Clin Exp Allergy. 2017 Apr;47(4):540-550. doi: 10.1111/cea.12862. Epub 2017 Jan 10. PMID 27883239